CLINICAL TRIAL: NCT06676020
Title: THE EFFECT OF THE TRAINING GIVEN TO THE PARENTS OF CHILDREN WITH FEBRILE CONVULSION WHO COME TO THE PAEDIATRIC EMERGENCY DEPARTMENT ON THE ANXIETY AND KNOWLEDGE LEVEL OF THE PARENTS
Brief Title: Effect of Febrile Convulsion Training on Anxiety and Knowledge
Acronym: FKT
Status: Not yet recruiting | Type: Observational
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Tugba KARAKUS TURKER, assistant professor, Uskudar University
Other Study IDs: UskudarUU
Record Dates: First submitted 2024-10-31; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Febrile Convulsion
Keywords: Febrile convulsion; EDUCATION; anxiety; knowledge level
MeSH Terms: conditions — Seizures, Febrile; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Febrile Convulsion Group
- Control Group

SUMMARY:
The research will be conducted to determine the effect of the training given to parents/caregivers on their knowledge, attitudes, practices and anxiety towards preventing febrile seizures in children. The research will be carried out as a randomised controlled experimental design in the Pediatric Emergency Department of Zeynep Kamil Women's and Children's Diseases Training and Research Hospital between October 2024 and October 2025.

DETAILED DESCRIPTION:
INTRODUCTION Febrile convulsion (FC) is defined as a type of seizure with fever in the absence of any 6 months to 5 years of age and is the most common neurological disorder of infants and young children. Although FC occurs in 2-4% of the entire paediatric population, 90% of cases occur between 6 months and 3 months of age. Simple FCs, defined as generalised seizures lasting less than 15 minutes, and represent the majority of febrile convulsions that do not recur within 24 hours. The risk of mortality and morbidity in FC is very low and there is no detectable brain damage associated with the disease. Complications of febrile seizures in children include psychosocial effects, cognitive deficits, hospital bed occupancy, prolonged hospitalisation and increased healthcare costs. In a 12-year follow-up of neurological complications from febrile seizures, delayed neurological development and abnormalities were found in 20% of children, neurological deficits in 10% and learning disabilities in 5%. Simple measures such as controlling fever, washing feet and using antipyretics can prevent the incidence of the disease and febrile seizure complications in children. Due to the concurrent relatively high prevalence of this disease in children, the occurrence of two important phenomena, such as fever and seizures, causes severe anxiety to parents and may impair the quality of life of the family. Informing parents by providing adequate knowledge and awareness about fever and seizures is an important step in reducing anxieties and worries. In a study conducted by Sheringham on 154 parents with children in febrile seizures, 54.3% of individuals receiving training had appropriate knowledge and there was a direct correlation between parents' knowledge and practice. In Flury's study, 91% of parents experienced severe anxiety when faced with febrile seizures, and the intensity of anxiety was significantly higher in untrained individuals than in trained individuals. Parmer, in a study of 140 parents with children who had febrile seizures in India, noted that 59.3% of parents were not aware of this disease and only 20% knew the normal values of body temperature. Education of parents was emphasised in the study. In the literature, the number of studies aiming to determine the level of knowledge by providing education to families of children hospitalised with FC is insufficient. Therefore, in the light of the literature, the study will be conducted to determine the impact of education given to parents/carers due to their knowledge, attitudes, practices and concerns in the prevention of febrile seizures in children.

ELIGIBILITY:
Inclusion Criteria:

1. Referral to paediatric emergency department with febrile convulsion
2. Children aged between 6 months and 5 years
3. Voluntary participation of the child and his/her family in the study.

Exclusion Criteria:

-

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The population of the study consisted of all children who applied to the Pediatric Emergency Department of Zeynep Kamil Women's and Children's Diseases Training and Research Hospital between October 2024 and October 2025. The sample of the study consisted of 66 parents.
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HAD) | one year
  Hospital Anxiety and Depression Scale (HAD) The scale is a four-point Likert-type assessment tool, and the scores of its items range from 0 to 3. However, each item is scored differently; items 1, 3, 5, 6, 8, 10, 11, and 13 show decreasing severity and are scored as 3, 2, 1, 0. On the other hand, items 2, 4, 7, 9, 12, and 14 are scored as 0, 1, 2, 3. The total scores of the subscales are obtained by adding the scores of these items. For the anxiety subscale, items 1, 3, 5, 7, 9, 11 and 13 are added; for the depression subscale, items 2, 4, 6, 8, 10, 12 and 14 are added.
Febrile Convulsion Knowledge Scale | one year
  Febrile Convulsion Knowledge Scale for Parents/Caregivers: In the febrile convulsion knowledge scale, items 1 and 4 are correct statements and the other items are incorrect statements. Incorrect statements should be reversed and calculated when scoring. The total score of the scale varies between 8 and 40, and higher scores indicate that parents/caregivers have more knowledge about febrile convulsions.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang MC, Huang CC, Thomas K. Febrile convulsions: development and validation of a questionnaire to measure parental knowledge, attitudes, concerns and practices. J Formos Med Assoc. 2006 Jan;105(1):38-48. doi: 10.1016/S0929-6646(09)60107-8. PMID 16440069
- [Background] Jones T, Jacobsen SJ. Childhood febrile seizures: overview and implications. Int J Med Sci. 2007 Apr 7;4(2):110-4. doi: 10.7150/ijms.4.110. PMID 17479160
- [Background] MacDonald BK, Johnson AL, Sander JW, Shorvon SD. Febrile convulsions in 220 children--neurological sequelae at 12 years follow-up. Eur Neurol. 1999;41(4):179-86. doi: 10.1159/000008048. PMID 10343147
- [Background] Verity CM, Greenwood R, Golding J. Long-term intellectual and behavioral outcomes of children with febrile convulsions. N Engl J Med. 1998 Jun 11;338(24):1723-8. doi: 10.1056/NEJM199806113382403. PMID 9624192
- [Background] Mohsen S, Mahboobeh SH: The effect of education based on health belief model (HBM) in mothers about behaviour of prevention from febrile convulsion in children. World J Med Sci. 2013, 9:30-5. 10.5829/idosi.wjms.2013.9.1.7617